CLINICAL TRIAL: NCT01798524
Title: An Observation Cohort Study of Kidney Allograft Recipients in England by Data Linkage Analysis
Brief Title: Kidney Allograft Recipients in England - an Observational Cohort Study
Acronym: KARE
Status: Completed | Type: Observational
Sponsor: University Hospital Birmingham NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Adnan Sharif, Dr, University Hospital Birmingham NHS Foundation Trust
Other Study IDs: HES-ONS
Record Dates: First submitted 2013-02-21; First posted 2013-02-26 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Kidney Transplantation
Keywords: Transplant; Kidney; England

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney allograft recipients

SUMMARY:
Kidney transplantation is the renal replacement therapy of choice for the majority of patients with end-stage kidney disease. Epidemiological studies of kidney allograft recipients can aid in the understanding of cause and effect of health and disease post-transplantation. The combination of health care and information technology has made the potential of transplant professionals to use health information effectively crucial to guide kidney transplant management. The aim of this study is to undertake an observational cohort study of kidney allograft recipients, supported by linking analysis across different database sources, to provide a comprehensive biomedical dataset of information.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplant alone
* English Transplant centre
* All ages
* Kidney allograft receipt between April 2001 and March 2012

Exclusion Criteria:

* Multiple organ transplant
* Transplant performed at non-English centre

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All kidney allograft recipients transplanted at an English transplant centre between April 2001 and March 2012
Sampling Method: Non-Probability Sample
Enrollment: 19688 (Actual)
Dates: Start 2011-11; Primary Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Mortality within the first year post kidney transplantation | One year

SECONDARY OUTCOMES:
Mortality beyond the first year post kidney transplantation | Up to 12 years

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Birmingham NHS Foundation trust, Birmingham, United Kingdom